CLINICAL TRIAL: NCT06776601
Title: Digital Therapy in Self-management of Chronic Obstructive Pulmonary Disease Patients：A Prospective, Open-labled, Multicenter Randomized Controlled Clinical Study.
Brief Title: Digital Therapy in Self-management of COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hongtao Niu, PhD, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ZRJY2023-QM16
Record Dates: First submitted 2024-12-21; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; adherence; inhaled medication; self management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital therapy intervention group (Experimental): Patients will receive individualized inhalation skills guidance after being tested by inhalation capacity measuring device, and be equipped with electronic inhalation monitoring devices, which can record their medication using data, reminding patients to use the medication on time, and correct their inhalation mistake. They can also check their inhalation record on their mobile phones. Clinicians can check the record every month to assess their adherence.
  Interventions: Behavioral: Full process digital therapy intervention package
- General management group (No Intervention): Patients will accept regular inhaler medication direction, and equipped with electronic inhalation monitoring that can only record medication using data.

INTERVENTIONS:
Behavioral: Full process digital therapy intervention package — Patients will receive individualized inhalation skills guidance after being tested by inhalation capacity measuring device, and be equipped with electronic inhalation monitoring devices, which can record their medication using data, reminding patients to use the medication on time, and correct their inhalation mistake. They can also check their inhalation record on their mobile phones. Clinicians can check the record every month to assess their adherence.
  Arms: Digital therapy intervention group

SUMMARY:
This project adopts a whole-process digital therapy intervention package composed of an inhalation technique assessment device, an electronic inhalant medication monitoring device and digital software to guide patients use the inhaler correctly personalizedly, record and manage the behavior data of chronic obstructive pulmonary disease (COPD) patients during the use of inhalant medication, and provide personalized reminders and feedback to patients according to the data. The purpose is to analyze whether this digital intervention scheme can reduce the number of acute exacerbations of COPD, improve the management effect of COPD, and reduce the burden of disease by improving the medication compliance of COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with COPD
2. Aged 40 and above
3. Had one or more severe acute exacerbations in the past year, and be in stable condition for the last 4 weeks
4. Can operate a smartphone proficiently
5. Take inhalation medication suits for the inhalation monitoring device as treatment
6. Fully understand and be willing to sign the informed consent form

Exclusion Criteria:

1. Certain comorbidities (e.g. unstable coronary complications)
2. Undergone thoracic, abdominal or ophthalmic surgery in recent 3 months
3. Pregnant or lactating women
4. ABS allergy history

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-09-18 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
severe exacerbation | 12 month
  Proportion of patients with severe acute exacerbation of COPD pulmonary disease during the follow-up period.

SECONDARY OUTCOMES:
First Second Forced Expiratory Volume/ Forced Vital Capacity | 12 month
  First Second Forced Expiratory Volume/Forced Vital Capacity (FEV1/FVC) measured by pulmonomete, %
First Second Forced Expiratory Volume percentage of estimated | 12 month
  First Second Forced Expiratory Volume (FEV1) percentage of estimated measured by pulmonomete, %
peak expiratory flow | 12 month
  peak expiratory flow (PEF) measured by pulmonomete, L/min
COPD Assessment Test score | 12 month
  COPD assessment test (CAT) is an eight-item questionnaire range from 0 to 40. Higher scroe represents heavier symptom.
modified Medical Research Council scale | 12 month
  The modified Medical Research Council (mMRC) scale stands for the level of patient self-report dyspnea. 0 is the minimum and 4 is the maximum.
St. George's Respiratory Questionnairefor chronic obstructive pulmonary disease (SGRQ) score | 12 month
  the SGRQ scroe range from 0 to 100. 0 represents for the least and 100represents for the most.
peak inspiratory flow rate | 12 month
  peak inspiratory flow rate (PIFR) measured by the sensor in the study
mild and moderate exacerbation | 12 month
  Proportion of patients with mild and moderate acute exacerbation of COPD pulmonary disease during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Hongtao Niu, PhD, Principal Investigator — China Japan Friendshi Hospital
Locations (1):
- China Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No